CLINICAL TRIAL: NCT02592824
Title: Phase III Study of Metabolic Intervention With Glutamate in Coronary Surgery II
Brief Title: Glutamate for Metabolic Intervention in Coronary Surgery II
Acronym: GLUTAMICSII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Region Örebro County (Other); University Hospital, Umeå (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Rolf Svedjeholm, Professor, MD, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT 2011-006241-15; Dnr 5.1-2015-77379 (Other: Swedish Medical Product Agency)
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Bypass Surgery; Postoperative Complications; Heart Failure
Keywords: glutamate, heart failure, coronary artery bypass surgery
MeSH Terms: conditions — Postoperative Complications; Heart Failure | interventions — Glutamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous glutamate infusion (Active Comparator): Intravenous infusion of 0.125M L-glutamic acid solution at a rate of 1.65 ml/kg BW and hour commencing at or up to 20 minutes before the release of aortic cross-clamp. The infusion is continued for two hours after declamping the aorta after which an additional 50 ml is given at a halved infusion rate.
  Interventions: Drug: glutamate infusion
- Intravenous saline infusion (Placebo Comparator): Intravenous infusion of saline at a rate of 1.65 ml/kg BW and hour commencing at or up to 20 minutes before the release of aortic cross-clamp. The infusion is continued for two hours after declamping the aorta after which an additional 50 ml is given at a halved infusion rate.
  Interventions: Drug: saline infusion

INTERVENTIONS:
Drug: glutamate infusion — Intravenous infusion of 0.125M L-glutamic acid solution at a rate of 1.65 ml/kg BW and hour commencing at or up to 20 minutes before the release of aortic cross-clamp. The infusion is continued for two hours after declamping the aorta after which an additional 50 ml is given at a halved infusion rate.
  Other Names: glutamate
  Arms: Intravenous glutamate infusion
Drug: saline infusion — Intravenous infusion of saline at a rate of 1.65 ml/kg BW and hour commencing at or up to 20 minutes before the release of aortic cross-clamp. The infusion is continued for two hours after declamping the aorta after which an additional 50 ml is given at a halved infusion rate.
  Other Names: saline
  Arms: Intravenous saline infusion

SUMMARY:
The aim of GLUTAMICS II is to evaluate whether intravenous glutamate infusion surgery reduces the risk of postoperative heart failure as measured by plasma NT-proBNP in patients undergoing moderate to high-risk coronary artery bypass graft surgery. Patients accepted for coronary artery bypass surgery of at least two vessel disease or left main stenosis with or without concomitant procedure and considered to be at moderate to high surgical risk preoperatively with regard to postoperative heart failure will be studied. The primary endpoint is postoperative increase of NT-proBNP from the day before surgery to the third postoperative day.

DETAILED DESCRIPTION:
In spite of the progress in cardiac surgery and perioperative management postoperative heart failure remains the leading cause of death and organ failure. Although acknowledged as a major problem in cardiac surgery there are no generally accepted criteria for the diagnosis of postoperative heart failure. This in turn could explain why treatment for postoperative heart failure is poorly documented with regard to clinical outcome.

Ischemia prior to cardiopulmonary bypass is the main cause of myocardial infarction after CABG. Available data demonstrate that ischemia and evolving myocardial infarction account for a large proportion of patients with postoperative heart failure after CABG.

Conventional treatment of postoperative heart failure presents a therapeutic dilemma as inotropic drugs not only aggravate ischemia and increase the size of evolving myocardial infarction, but also stimulate apoptotic processes that may have adverse long-term consequences.

The role of inotropes in cardiac surgery is therefore controversial. Some authors claim that liberal use of inotropes and goal-directed haemodynamic therapy can improve outcome whereas other report that liberal use of inotropes is associated with increased morbidity and mortality.

Alternative measures that can enhance myocardial recovery and function without putting further strain on the heart are therefore desirable.

Glutamate could influence outcome after myocardial ischemia by two different biochemical mechanisms. First, glutamate improves myocardial tolerance to ischemia by facilitated anaerobic metabolism and substrate level phosphorylation during ischemia. The second mechanism is related to the anaplerotic role of glutamate. Glutamate plays a key role for replenishment of Krebs cycle intermediates lost during ischemia, which enhances post-ischemic recovery of myocardial oxidative metabolism and function.

Promoting metabolic and functional recovery with metabolic support represents a novel concept in the treatment of heart failure after acute ischemia. Animal experiments suggest that glutamate increases myocardial tolerance to ischemia and that glutamate promotes post-ischemic recovery. Intravenous glutamate improved metabolic and hemodynamic recovery in humans early after CABG. Early clinical experience with intravenous metabolic support showed that the need for inotropes could be substantially reduced while clinical outcomes with regard to postoperative mortality, postoperative renal dysfunction and long-term survival compared favourably with the literature. This encouraging experience contributed to the initiation of the first GLUTAMICS-trial.

The first GLUTAMICS-trial investigated if intravenous glutamate infusion given in association with surgery for acute coronary syndrome could prevent myocardial injury, postoperative heart failure and reduce mortality. The study was negative with regard to the primary endpoint, which was a composite of postoperative mortality, perioperative myocardial infarction and left ventricular failure at weaning from cardiopulmonary bypass.

However, the study included a high proportion of low risk patients. Furthermore, the design of the primary endpoint suffered from liberal preemptive use of inotropes in patients anticipated to have weaning problems. It became evident at clinical endpoint committee meetings that preemptive use of inotropes prevented detection of weaning problems in patients who later developed severe heart failure. The secondary endpoint severe circulatory failure discriminated mild short-lasting heart failure at weaning from cardiopulmonary bypass from clinically significant heart failure requiring substantial circulatory support and leading to prolonged ICU stay or death. In the glutamate treated patients the relative risk of developing severe circulatory failure was reduced by more than 50% in most risk groups undergoing isolated CABG.

The first GLUTAMICS trial also included a substudy consisting of a blinded evaluation of NT-proBNP as a marker for postoperative heart failure.

Due to the lack of generally accepted criteria for postoperative heart failure, the evaluation of treatment is difficult. Consequently, comparative studies on different treatment strategies of heart failure after cardiac surgery are sparse given the magnitude of the problem.

Natriuretic peptides have been extensively studied in cardiology. In patients with chronic heart failure markedly increased BNP and NT-pro BNP levels are associated with poor prognosis. The response of natriuretic peptides to heart failure treatment has significant prognostic implications, and non-responders have a poor prognosis.

In cardiac surgery NT-proBNP increase was more pronounced in patients requiring inotropes. High postoperative levels of BNP and NT-proBNP were associated with worse outcome, both in the short- and long-term.

The first GLUTAMICS-trial permitted a blinded prospective evaluation of NT-proBNP by a clinical end-points committee relying on strict prespecified criteria with regard to postoperative heart failure. Data to be published demonstrate that postoperative NT-proBNP (day 1 and day 3) levels were strong predictors for severe heart failure associated with extended ICU stay or death. This implies that postoperative NT-proBNP could serve as a measure to assess efficacy of treatment and preventive strategies for postoperative heart failure. Albeit, a surrogate marker for postoperative heart failure it provides the advantage of a standardized and objective analysis, which makes the study reproducible.

AIM

The aim is to confirm findings in subgroups from the first GLUTAMICS-trial that intravenous glutamate infusion reduces the risk of postoperative heart failure in moderate to high risk patients undergoing coronary artery surgery by showing a reduced increase of NT-proBNP postoperatively.

PATIENTS

Patients accepted for coronary artery bypass surgery of at least two vessel disease or left main stenosis with or without concomitant procedure considered to be at moderate to high surgical risk preoperatively with regard to postoperative heart failure.

310 patients are planned to be included after informed written consent.

Exclusion criteria: patients with ambiguous food allergies that trigger shortness of breath, headache or flushing; patients> 85 years, previous cardiac surgery, patients who are in such bad condition that they cannot be asked to participate, patients who for linguistic or other reasons are unable to provide informed consent, severe renal failure with preoperative dialysis or calculated GFR <30 mL / min, patients requiring inotropic drugs or mechanical circulatory support (intra-aortic balloon pump) due to circulatory failure even before they enrolled in the study, patients who undergo surgery without the heart-lung machine (off-pump), patients who undergo concomitant Maze-procedure or surgery of ascending aorta.

STUDY DESIGN

The GLUTAMICS II is an investigator initiated prospective, randomized, placebo controlled, double-blind trial with parallel assignment to glutamate or placebo (saline). The trial is externally randomized and randomization is stratified for patients undergoing isolated CABG and for those having CABG with concomitant procedure.

INTERVENTION

Patients are randomly allocated to blinded intravenous infusion of 0.125M L-glutamic acid solution or saline at a rate of 1.65 ml/kg and hour commencing at or up to 20 minutes before the release of aortic cross-clamp. The infusion is continued for two hours after declamping the aorta after which an additional 50 ml is given at a halved infusion rate.

PRIMARY ENDPOINT

The primary endpoint is a postoperative increase of NT-proBNP from the day before surgery to the third postoperative day.

SECONDARY ENDPOINTS

Secondary endpoints are the absolute postoperative plasma levels of NT-proBNP day 1 and day 3.

SAFETY VARIABLES

Postoperative mortality (30 days + hospitals), stroke within 24 hours and SUSARs

SAMPLE SIZE

Sample size is based on available results from the first GLUTAMICS study. In that study, the following increase of NT-proBNP from the preoperative value to third postoperative day (mean ± SD) were observed in patients with LVEF ≤ 0.30 or EuroSCORE II ≥ 3.0 undergoing coronary artery surgery for with or without concomitant procedure.

Glutamate (n=71): 5261 ± 4409

Placebo (n=62): 7112 ± 6454

Sample size assessment by external statistical expertise (80% power, 5% risk level; two-sided test) suggests 141 patients in each group. To account for failed sampling and other loss we plan a total of 310 patients.

INTERIM ANALYSIS

Interim analysis will be performed by an external independent statistician after 160 patients by an adaptive design as reported in detail to the Swedish Medical Product Agency.

Update August 30, 2020: Interim analysis in December 2017 supported the original sample size assessment and the aim was set to reach 300 patients with complete data for the primary endpoint. The original goal of 280 patients with complete data has been reached and the study is approaching 300 but as study solutions will expire September 30, 2020 this will be the last date for inclusion of patients into the trial.

ETHICAL CONSIDERATIONS

A concern with the use of glutamate is that it may act as an excitotoxin under certain conditions and participate in events leading to neurological damage. However, brain tissue concentrations of glutamate are more than fifty-fold higher than in blood whereas the dosage used only elevates blood levels three-fold. Neurological outcome has been carefully monitored when intravenous infusions have been used in clinical practice without evidence of adverse effects. No evidence of subclinical neurological injury associated with intravenous glutamate infusion could be detected by the S-100B measurements and no differences in neurological outcome or other adverse events were found in the GLUTAMICS trial.

After written informed consent eligible patients will be enrolled in the study. The study will be performed according to the Helsinki Declaration of Human Rights and is approved by the Regional Ethical Review Board in Linköping (Dnr 2011/498-31; Dnr 2015/333-32).

The Swedish Medical Products Agency requests surveillance and unblinding in cases of CT-verified stroke within 24 hours of surgery, mortality and suspected unexpected serious adverse reactions (SUSAR). External monitoring of all key data, written informed consent and unblinding procedures will be done.

ELIGIBILITY:
Inclusion Criteria:

Patients accepted for coronary artery bypass surgery of at least two vessel disease or left main stenosis with or without concomitant procedure considered to be at moderate to high surgical risk preoperatively with regard to postoperative heart failure due to:

• EuroSCORE II ≥ 3.0 with at least one of the following cardiac or procedure related risk factors:

* LVEF ≤ 0.50
* CCS class IV
* Recent Myocardial Infarct (≤ 90 days)
* Emergency / Urgent procedure (as defined in EuroSCORE II)
* CABG with aortic or mitral valve procedure

OR

• LVEF ≤ 0.30 regardless of EuroSCORE II

Exclusion Criteria:

* age > 85 years
* ambiguous food allergies that trigger shortness of breath, headache or flushing
* previous cardiac surgery
* patients who are in such bad condition that they cannot be asked to participate
* patients who because of linguistic or other reasons are unable to provide informed consent
* severe renal failure with preoperative dialysis or calculated GFR <30 mL / min
* patients requiring mechanical circulatory support (intra-aortic balloon pump) due to circulatory failure before they are enrolled in the study
* surgery without heart-lung machine (off-pump)
* concomitant Maze-procedure
* surgery of ascending aorta
* surgery of both aortic and mitral valve

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Svedjeholm, Professor, Study Chair — University Hospital, Linkoeping; Farkas Vanky, MD, PhD, Principal Investigator — University Hospital, Linkoeping
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - University Hospital Linköping, Linköping
  - University Hospital Örebro, Örebro
  - University Hospital Umeå, Umeå

REFERENCES:
- [Background] O'Connor GT, Birkmeyer JD, Dacey LJ, Quinton HB, Marrin CA, Birkmeyer NJ, Morton JR, Leavitt BJ, Maloney CT, Hernandez F, Clough RA, Nugent WC, Olmstead EM, Charlesworth DC, Plume SK. Results of a regional study of modes of death associated with coronary artery bypass grafting. Northern New England Cardiovascular Disease Study Group. Ann Thorac Surg. 1998 Oct;66(4):1323-8. doi: 10.1016/s0003-4975(98)00762-0. PMID 9800828
- [Background] Fellahi JL, Parienti JJ, Hanouz JL, Plaud B, Riou B, Ouattara A. Perioperative use of dobutamine in cardiac surgery and adverse cardiac outcome: propensity-adjusted analyses. Anesthesiology. 2008 Jun;108(6):979-87. doi: 10.1097/ALN.0b013e318173026f. PMID 18497597
- [Background] Gillies M, Bellomo R, Doolan L, Buxton B. Bench-to-bedside review: Inotropic drug therapy after adult cardiac surgery -- a systematic literature review. Crit Care. 2005 Jun;9(3):266-79. doi: 10.1186/cc3024. Epub 2004 Dec 16. PMID 15987381
- [Background] Mebazaa A, Pitsis AA, Rudiger A, Toller W, Longrois D, Ricksten SE, Bobek I, De Hert S, Wieselthaler G, Schirmer U, von Segesser LK, Sander M, Poldermans D, Ranucci M, Karpati PC, Wouters P, Seeberger M, Schmid ER, Weder W, Follath F. Clinical review: practical recommendations on the management of perioperative heart failure in cardiac surgery. Crit Care. 2010;14(2):201. doi: 10.1186/cc8153. Epub 2010 Apr 28. PMID 20497611
- [Background] Slogoff S, Keats AS. Does perioperative myocardial ischemia lead to postoperative myocardial infarction? Anesthesiology. 1985 Feb;62(2):107-14. doi: 10.1097/00000542-198502000-00002. PMID 3970360
- [Background] Vanky F, Hakanson E, Maros T, Svedjeholm R. Different characteristics of postoperative heart failure after surgery for aortic stenosis and coronary disease. Scand Cardiovasc J. 2004 Jun;38(3):152-8. doi: 10.1080/14017430410029734. PMID 15223713
- [Background] Vanky FB, Hakanson E, Svedjeholm R. Long-term consequences of postoperative heart failure after surgery for aortic stenosis compared with coronary surgery. Ann Thorac Surg. 2007 Jun;83(6):2036-43. doi: 10.1016/j.athoracsur.2007.01.031. PMID 17532392
- [Background] Dahlin LG, Olin C, Svedjeholm R. Perioperative myocardial infarction in cardiac surgery--risk factors and consequences. A case control study. Scand Cardiovasc J. 2000 Oct;34(5):522-7. doi: 10.1080/140174300750064710. PMID 11191945
- [Background] Khoynezhad A, Jalali Z, Tortolani AJ. Apoptosis: pathophysiology and therapeutic implications for the cardiac surgeon. Ann Thorac Surg. 2004 Sep;78(3):1109-18. doi: 10.1016/j.athoracsur.2003.06.034. PMID 15337071
- [Background] Maroko PR, Kjekshus JK, Sobel BE, Watanabe T, Covell JW, Ross J Jr, Braunwald E. Factors influencing infarct size following experimental coronary artery occlusions. Circulation. 1971 Jan;43(1):67-82. doi: 10.1161/01.cir.43.1.67. No abstract available. PMID 5540853
- [Background] Lazar HL, Buckberg GD, Foglia RP, Manganaro AJ, Maloney JV Jr. Detrimental effects of premature use of inotropic drugs to discontinue cardiopulmonary bypass. J Thorac Cardiovasc Surg. 1981 Jul;82(1):18-25. PMID 7242127
- [Background] Thackray S, Easthaugh J, Freemantle N, Cleland JG. The effectiveness and relative effectiveness of intravenous inotropic drugs acting through the adrenergic pathway in patients with heart failure-a meta-regression analysis. Eur J Heart Fail. 2002 Aug;4(4):515-29. doi: 10.1016/s1388-9842(02)00041-7. PMID 12167393
- [Background] Aya HD, Cecconi M, Hamilton M, Rhodes A. Goal-directed therapy in cardiac surgery: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):510-7. doi: 10.1093/bja/aet020. Epub 2013 Feb 27. PMID 23447502
- [Background] Giglio M, Dalfino L, Puntillo F, Rubino G, Marucci M, Brienza N. Haemodynamic goal-directed therapy in cardiac and vascular surgery. A systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2012 Nov;15(5):878-87. doi: 10.1093/icvts/ivs323. Epub 2012 Jul 24. PMID 22833509
- [Background] Shahin J, DeVarennes B, Tse CW, Amarica DA, Dial S. The relationship between inotrope exposure, six-hour postoperative physiological variables, hospital mortality and renal dysfunction in patients undergoing cardiac surgery. Crit Care. 2011 Jul 7;15(4):R162. doi: 10.1186/cc10302. PMID 21736726
- [Background] Lazar HL, Buckberg GD, Manganaro AJ, Becker H, Maloney JV Jr. Reversal of ischemic damage with amino acid substrate enhancement during reperfusion. Surgery. 1980 Nov;88(5):702-9. PMID 7434210
- [Background] Pisarenko OI. Mechanisms of myocardial protection by amino acids: facts and hypotheses. Clin Exp Pharmacol Physiol. 1996 Aug;23(8):627-33. doi: 10.1111/j.1440-1681.1996.tb01748.x. PMID 8886480
- [Background] Rau EE, Shine KI, Gervais A, Douglas AM, Amos EC 3rd. Enhanced mechanical recovery of anoxic and ischemic myocardium by amino acid perfusion. Am J Physiol. 1979 Jun;236(6):H873-9. doi: 10.1152/ajpheart.1979.236.6.H873. No abstract available. PMID 443452
- [Background] Safer B. The Metabolic Significance of the Malate-Aspartate Cycle in Heart. Circ Res. 1975 Nov;37(5):527-33. doi: 10.1161/01.res.37.5.527. No abstract available. PMID 172258
- [Background] Peuhkurinen KJ. Regulation of the tricarboxylic acid cycle pool size in heart muscle. J Mol Cell Cardiol. 1984 Jun;16(6):487-95. doi: 10.1016/s0022-2828(84)80637-9. PMID 6748086
- [Background] Pisarenko OI, Novikova EB, Serebryakova LI, Tskitishvili OV, Ivanov VE, Studneva IM. Function and metabolism of dog heart in ischemia and in subsequent reperfusion: effect of exogenous glutamic acid. Pflugers Arch. 1985 Dec;405(4):377-83. doi: 10.1007/BF00595691. PMID 2867519
- [Background] Haas GS, DeBoer LW, O'Keefe DD, Bodenhamer RM, Geffin GA, Drop LJ, Teplick RS, Daggett WM. Reduction of postischemic myocardial dysfunction by substrate repletion during reperfusion. Circulation. 1984 Sep;70(3 Pt 2):I65-74. PMID 6430593
- [Background] Engelman RM, Rousou JA, Flack JE 3rd, Iyengar J, Kimura Y, Das DK. Reduction of infarct size by systemic amino acid supplementation during reperfusion. J Thorac Cardiovasc Surg. 1991 May;101(5):855-9. PMID 1673733
- [Background] Pisarenko OI, Lepilin MG, Ivanov VE. Cardiac metabolism and performance during L-glutamic acid infusion in postoperative cardiac failure. Clin Sci (Lond). 1986 Jan;70(1):7-12. doi: 10.1042/cs0700007. PMID 2867848
- [Background] Svedjeholm R, Vanhanen I, Hakanson E, Joachimsson PO, Jorfeldt L, Nilsson L. Metabolic and hemodynamic effects of intravenous glutamate infusion early after coronary operations. J Thorac Cardiovasc Surg. 1996 Dec;112(6):1468-77. doi: 10.1016/S0022-5223(96)70005-3. PMID 8975838
- [Background] Svedjeholm R, Huljebrant I, Hakanson E, Vanhanen I. Glutamate and high-dose glucose-insulin-potassium (GIK) in the treatment of severe cardiac failure after cardiac operations. Ann Thorac Surg. 1995 Feb;59(2 Suppl):S23-30. doi: 10.1016/0003-4975(94)00918-w. PMID 7840695
- [Background] Svedjeholm R, Vidlund M, Vanhanen I, Hakanson E. A metabolic protective strategy could improve long-term survival in patients with LV-dysfunction undergoing CABG. Scand Cardiovasc J. 2010 Feb;44(1):45-58. doi: 10.3109/14017430903531008. PMID 20141344
- [Background] Vidlund M, Hakanson E, Friberg O, Juhl-Andersen S, Holm J, Vanky F, Sunnermalm L, Borg JO, Sharma R, Svedjeholm R. GLUTAMICS--a randomized clinical trial on glutamate infusion in 861 patients undergoing surgery for acute coronary syndrome. J Thorac Cardiovasc Surg. 2012 Oct;144(4):922-930.e7. doi: 10.1016/j.jtcvs.2012.05.066. Epub 2012 Jun 19. PMID 22721612
- [Background] de Lemos JA, McGuire DK, Drazner MH. B-type natriuretic peptide in cardiovascular disease. Lancet. 2003 Jul 26;362(9380):316-22. doi: 10.1016/S0140-6736(03)13976-1. PMID 12892964
- [Background] Karlstrom P, Alehagen U, Boman K, Dahlstrom U; UPSTEP-study group. Brain natriuretic peptide-guided treatment does not improve morbidity and mortality in extensively treated patients with chronic heart failure: responders to treatment have a significantly better outcome. Eur J Heart Fail. 2011 Oct;13(10):1096-103. doi: 10.1093/eurjhf/hfr078. Epub 2011 Jun 29. PMID 21715446
- [Background] Reyes G, Fores G, Rodriguez-Abella RH, Cuerpo G, Vallejo JL, Romero C, Pinto A. NT-proBNP in cardiac surgery: a new tool for the management of our patients? Interact Cardiovasc Thorac Surg. 2005 Jun;4(3):242-7. doi: 10.1510/icvts.2004.101576. Epub 2005 Mar 30. PMID 17670401
- [Background] Nozohoor S, Nilsson J, Algotsson L, Sjogren J. Postoperative increase in B-type natriuretic peptide levels predicts adverse outcome after cardiac surgery. J Cardiothorac Vasc Anesth. 2011 Jun;25(3):469-75. doi: 10.1053/j.jvca.2010.07.002. Epub 2010 Sep 9. PMID 20829070
- [Background] Fox AA, Nascimben L, Body SC, Collard CD, Mitani AA, Liu KY, Muehlschlegel JD, Shernan SK, Marcantonio ER. Increased perioperative b-type natriuretic peptide associates with heart failure hospitalization or heart failure death after coronary artery bypass graft surgery. Anesthesiology. 2013 Aug;119(2):284-94. doi: 10.1097/ALN.0b013e318299969c. PMID 23695172
- [Derived] Holm J, Vanky F, Svedjeholm R. Association of Glutamate Infusion With Risk of Acute Kidney Injury After Coronary Artery Bypass Surgery: A Pooled Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2024 Jan 2;7(1):e2351743. doi: 10.1001/jamanetworkopen.2023.51743. PMID 38252440
- [Derived] Holm J, Vanky F, Svedjeholm R. Glutamate Infusion Reduces Myocardial Dysfunction after Coronary Artery Bypass Grafting According to NT-proBNP: Summary of 2 Randomized Controlled Trials (GLUTAmate for Metabolic Intervention in Coronary Surgery [GLUTAMICS I-II]). Am J Clin Nutr. 2023 Nov;118(5):930-937. doi: 10.1016/j.ajcnut.2023.08.012. Epub 2023 Aug 30. PMID 37657522
- [Derived] Holm J, Ferrari G, Holmgren A, Vanky F, Friberg O, Vidlund M, Svedjeholm R. Effect of glutamate infusion on NT-proBNP after coronary artery bypass grafting in high-risk patients (GLUTAMICS II): A randomized controlled trial. PLoS Med. 2022 May 9;19(5):e1003997. doi: 10.1371/journal.pmed.1003997. eCollection 2022 May. PMID 35533197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 321 patients gave written informed consent.
  7 patients were not randomized ( change of procedure n=2; forgetfulness n=5)
Period: Overall Study
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
Started | 155 (7 patients not completed (Intraoperative exclusion criteria n= 5; Lost CRF n=2)) | 159 (4 patients not completed ( Intraoperative exclusion criteria n=3; Lost CRF n=1))
Completed | 148 | 155
Not Completed | 7 | 4
Not completed — Protocol Violation | 5 | 3
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion | Total
Number analyzed (Participants) | 148 | 155 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (7) | 75 (7) | 74 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 79
  Male | 112 | 112 | 224
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 148 | 155 | 303
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 148 | 155 | 303
NTproBNP ng/L [Mean (Standard Deviation); unit: ng/L] | 2680 (4595) | 2354 (3124) | 2513 (3909)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Increase of Plasma NT-proBNP
Description: Postoperative increase of NT-proBNP reflects postoperative myocardial dysfunction sustained in association with surgery. NT-proBNP usually peaks on the third to fourth postoperative day after coronary artery bypass surgery.
  In the first GLUTAMICS trial a good agreement between hemodynamic criteria for postoperative heart failure and postoperative NT-proBNP was found.
Time Frame: from the day before surgery to the third postoperative day
Population: Incomlete sampling of NT-proBNP in the Glutamate infusion group (n=3) and Saline infusion group (n=5).
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
Number analyzed (Participants) | 145 | 150
ng/L | 5390 (5396) | 6452 (5215)
Statistical Analysis 1: Comparison: Intravenous Glutamate Infusion vs Intravenous Saline Infusion; Two-sided Student's t-test used for sample size estimation which was based on data from the first GLUTAMICS trial; Test type: Superiority; p = 0.086, t-test, 2 sided

2. Secondary Outcome: Postoperative Plasma Level of NT-proBNP
Description: Postoperative NT-proBNP reflects postoperative myocardial dysfunction.
Time Frame: first postoperative day
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
Number analyzed (Participants) | 148 | 153
ng/L | 4438 (4879) | 4420 (4236)
Statistical Analysis 1: Comparison: Intravenous Glutamate Infusion vs Intravenous Saline Infusion; Test type: Superiority; p = 0.97, t-test, 2 sided

3. Secondary Outcome: Postoperative Plasma Level of NT-proBNP
Description: Postoperative NT-proBNP reflects postoperative myocardial dysfunction.
Time Frame: third postoperative day
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
Number analyzed (Participants) | 145 | 150
ng/L | 8055 (7546) | 8804 (6606)
Statistical Analysis 1: Comparison: Intravenous Glutamate Infusion vs Intravenous Saline Infusion; Test type: Superiority; p = 0.36, t-test, 2 sided

4. Secondary Outcome: Number of Participants With Incidence of Stroke
Description: Postoperative stroke was defined as neurological or cognitive deficit with a cerebral injury verified on (Computed Tomography) CT-scan. All suspected cases of stroke underwent CT-scan.
  Stroke within 24 h of surgery was defined as a stroke that occurred within 24 h of surgery or signs of a stroke, when first assessable in deeply sedated patients on a ventilator.
Time Frame: within 24 hours from surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
Number analyzed (Participants) | 148 | 155
Participants | 0 | 4

5. Secondary Outcome: Incidence of Mortality
Description: Postoperative mortality was defined as mortality within 30 days of surgery.
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
Number analyzed (Participants) | 148 | 155
Participants | 1 | 6

6. Secondary Outcome: Incidence of Unexpected Adverse Events
Description: suspected unexpected serious adverse reaction
Time Frame: within 24 hours from infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
Number analyzed (Participants) | 148 | 155
Participants | 0 | 0

7. Other Pre Specified Outcome: Copeptin Substudy
Description: Exploratory assessment of plasma-Copeptin related to NT-proBNP
Time Frame: preoperative, first and third postoperative day
Reporting Status: Not Posted

8. Post Hoc Outcome: Postoperative Increase of Plasma NT-proBNP in Patients Without Diabetes
Description: Postoperative increase of NT-proBNP reflects postoperative myocardial dysfunction sustained in association with surgery. NT-proBNP usually peaks on the third to fourth postoperative day after coronary artery bypass surgery.
  Previous observations suggest a blunted effect of glutamate in diabetic hearts.
Time Frame: from preoperative level to the third postoperative day
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
Number analyzed (Participants) | 75 | 83
ng/L | 4503 (4846) | 6825 (5671)
Statistical Analysis 1: Comparison: Intravenous Glutamate Infusion vs Intravenous Saline Infusion; Test type: Superiority; p = 0.007, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events agree with clinicaltrials.gov definitions but are mainly related to the surgical procedure
Arm/Group | Intravenous Glutamate Infusion | Intravenous Saline Infusion
All-Cause Mortality (participants affected / at risk) | 1/148 | 6/155
Serious Adverse Events (participants affected / at risk) | 65/148 | 79/155
Other Adverse Events (participants affected / at risk) | 31/148 | 31/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Glutamate Infusion (N=148) | Intravenous Saline Infusion (N=155)
Postoperative Atrial Fibrillation (Surgical and medical procedures) | 31 | 39 — Postoperative atrial fibrillation associated with more than one weeks hospital stay at the cardiac surgical unit
Acute Kidney Injury (Surgical and medical procedures) | 26 | 40 — AKI defined as a postoperative increase of p-creatinine by at least 50% from preoperative level
Reoperation for bleeding (Surgical and medical procedures) | 11 | 17
Periperative myocardial injury (Surgical and medical procedures) | 20 | 18 — CK-MB on the first postoperative day > 70 ug/L or Troponin-T on postoperative day 3 > 2000 ng/L
Postoperative Stroke (Nervous system disorders) | 5 | 7 — Stroke during hospital stay. Postoperative stroke was defined as neurological or cognitive deficit with a cerebral injury verified on (Computed Tomography) CT-scan. All suspected cases of stroke underwent CT-scan.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Glutamate Infusion (N=148) | Intravenous Saline Infusion (N=155)
Postoperative Atrial fibrillation (Surgical and medical procedures) | 31 | 31 — Postoperative atrial fibrillation not associated with hospital stay at the cardiac surgical unit exceeding one week

LIMITATIONS AND CAVEATS:
The main limitations of the study are: (i) it relies on a surrogate marker for heart failure (ii) the proportion of patients with diabetes had almost doubled compared to the cohort used for the sample size estimation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02592824/Prot_SAP_000.pdf